CLINICAL TRIAL: NCT06704165
Title: Evaluation of Apical Root Resorption in Dental Deep Bite Correction by Twin Slot Orthodontic Bracket; a Clinical Trial Study
Brief Title: Evaluation of Apical Root Resorption in Dental Deep Bite Correction by Twin Slot Orthodontic Bracket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Alaa Abd Elsalam Ramadan Salama, Evaluation of Apical Root Resorption in Dental Deep Bite Correction by Twin Slot Orthodontic Bracket; A Clinical Trial Study, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-OR-22-02
Record Dates: First submitted 2024-11-18; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Volumetric Root Resorption
Keywords: intrusion,root resorption
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evaluate the possible apical root resorption by double slot bracket withwire in high level slot. (Experimental): Control group : patients will receive a conventional therapy with Double slot bracket with the wire in high level for the treatment of anterior deep bite .
  Interventions: Procedure: Orthodontic treatment using double slot bracket wire in high level slot
- Evaluate the possible apical root resorption by double slot bracket with wire in low level slot. (Experimental): investigational group will receives the new treatment therapy by using Double slot bracket with the wire in low level for the treatment of anterior deep bite .
  Interventions: Procedure: Orthodontic treatment using double slot bracket with wire in low level slot

INTERVENTIONS:
Procedure: Orthodontic treatment using double slot bracket wire in high level slot — patients will receives the new treatment therapy by using Double slot bracket with the wire in low level for the treatment of anterior deep bite .
  Arms: Evaluate the possible apical root resorption by double slot bracket withwire in high level slot.
Procedure: Orthodontic treatment using double slot bracket with wire in low level slot — patients will receives the new treatment therapy by using Double slot bracket with the wire in high level for the treatment of anterior deep bite .
  Arms: Evaluate the possible apical root resorption by double slot bracket with wire in low level slot.

SUMMARY:
Evaluate the possible apical root resorption during deep bite correction by double slot bracket with low level slot versus high level slot using CBCT.

DETAILED DESCRIPTION:
Group (A): Patients will be treated with double slot brackets using low level slot in deep bite correction. Group (B): Patients will be treated with double slot brackets using high level slot in deep bite correction.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients to avoid any sexual dimorphism which may affect the comparison.
2. Age range from 18 to 23year.
3. Patients with anterior dento alveolar deep bite.
4. Angle class I or class II malocclusion with minimal crowding.
5. Healthy compliant and motivated patient.
6. No missing of any tooth except wisdom teeth

Exclusion Criteria:

* 1. Previous orthodontic treatments. 2. Any systemic or bone diseases. 3. Pregnant and lactating patient. 4. Prosthetic replacement in lower anterior teeth. 5. periodontitis with pocket depth more than 5 mm

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | "through study completion, an average of 1 year".
  Evaluate and compare the amount of volumetric root resorption. CBCT used in volumetric image.

SECONDARY OUTCOMES:
Secondary Outcome Measure | "through study completion, an average of 1 year".
  Evaluation of alveolar bone changes using CBCT.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Abdo Ibrahim, professor, Principal Investigator — AL Azher university
Locations (1):
- Alaa Salama, Bohira, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No